CLINICAL TRIAL: NCT00124969
Title: Influence of Amlodipine on the Mortality of Patients With End-Stage Renal Failure (ADAM [Amlodipine and Dialysis Patients, Action on Mortality])
Brief Title: Influence of Amlodipine on the Mortality of Patients With End-Stage Renal Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADAM; AML-D-01-001G
Record Dates: First submitted 2005-06-30; First posted 2005-07-29 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2006-10

CONDITIONS: Kidney Failure, Chronic
Keywords: End-stage renal disease, hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Amlodipine
  Interventions: Drug: Amlodipine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amlodipine — 10mg
  Other Names: Placebo
  Arms: 1
Drug: Placebo — 10mg
  Arms: 2

SUMMARY:
Patients with end-stage renal failure have a markedly higher mortality because of cardiovascular events in comparison with the normal population. Disorders in the calcium metabolism, such as calcification of the vessel walls, occur very frequently. There are indications that calcium channel blockers are capable of lowering the cardiovascular mortality in patients with end-stage renal failure.

It is intended to carry out a prospective, randomized, double-blind, placebo-controlled, multicenter study in order to find out if the calcium channel blocker amlodipine is able to reduce the mortality of patients with end-stage renal failure.

The investigation will be carried out after suitable explanation and written informed consent in 356 patients aged between 18 and 90 years with end-stage renal failure and chronic haemodialysis treatment. The patients will be randomized to either treatment with amlodipine 10 mg/day or placebo. The occurrence of events will be documented and evaluated prospectively over a period of 30 months.

DETAILED DESCRIPTION:
Trial protocol for ADAM Study

1.1 General Data:

1. Title of the Study: Influence of Amlodipine on the Mortality of Patients with End-Stage Renal Failure (abbreviated title: ADAM [Amlodipine and Dialysis Patients, Action on Mortality])
2. Study Directors:

   Prof. Dr. med. Martin Tepel, Charite University of Berlin, Campus Benjamin Franklin, Medizinische Klinik IV, Hindenburgdamm 30, 12200 Berlin, Germany. Tel.: +49-30 8445 2305, Fax: +49-30 8445 4235, e-mail: Martin.Tepel@charite.de

   Statistics:

   PD Dr. rer. nat. Dr. med. Werner Th. Hopfenmüller, Charite University of Berlin, Campus Benjamin Franklin, Institut für Medizinische Statistik und Biometrie, Hindenburgdamm 30, 12200 Berlin, Germany. Tel.: +49-30 8445 3512 Fax: +49-30 8445 4471
3. Summary of the ADAM Study:

   Patients with end-stage renal failure have a markedly higher mortality because of cardiovascular events in comparison with the normal population. Disorders in the calcium metabolism, such as calcification of the vessel walls, occur very frequently. There are indications that calcium channel blockers are capable of lowering the cardiovascular mortality in patients with end-stage renal failure. It is intended to carry out a prospective, randomized, double-blind, placebo-controlled, multicenter study in order to find out if the calcium channel blocker amlodipine is able to reduce the mortality of patients with end-stage renal failure.

   The investigation will be carried out after suitable explanation and written informed consent in 356 patients aged between 18 and 90 years with end-stage renal failure and chronic haemodialysis treatment. The patients will be randomized to either treatment with amlodipine 10 mg/day or placebo. The occurrence of events will be documented and evaluated prospectively over a period of 30 months.
4. Sponsor:

   There is no sponsor for this study. The study was initiated by the study directors themselves. The Pfizer company (Karlsruhe) is supporting the project financially and materially.
5. Trial Center:

   It is planned to carry out the study in the Berlin/Brandenburg area and in North Rhine Westphalia. The doctors responsible in the respective Trial Centers will be notified to the Ethics Committee immediately after enrolment. At present there are no enrolled Trial Centers.
6. Ethics Committee:

   The present Trial Protocol has been presented to the Ethics Committee of the Free University of Berlin (chairman: Prof. Dr. med. D. Ganten) for review.
7. Other Ethics Committees:

   This Trial Protocol has so far not been presented to any other institutions for assessment.
8. Classification of the Study:

   This is a Phase IV study. The study will be carried out with a licensed medicament (amlodipine) with a licensed indication (hypertension). This is a clinical study in patients who are legally competent and who are capable of understanding the nature, importance and scope of the clinical trial.
9. Legal Basis German Medicines Act

1.2 Justification and Aim of the Study:

1. Aim and Hypothesis:

   The aim of the study is to show that the administration of the calcium antagonist amlodipine significantly reduces mortality in patients with end-stage renal failure.

   Hypothesis: Amlodipine reduces the mortality in patients with end-stage renal failure.
2. Current Status of Research and Basis for the Performance of the Study:

   The life expectancy of patients with end-stage renal failure is nowadays still less than 10 years. The annual mortality rate of patients with end-stage renal failure is almost 25%. Death of patients with end-stage renal failure is frequently the consequence of cardiovascular events. Cardiovascular events in patients with dialysis-dependent renal failure are particularly frequently seen because the traditional risk factors, such as diabetes, hypertension, hyperlipidemia and smoking, are frequently present in this group. In addition, there are also numerous risk factors associated with the renal failure, such as increased oxidative stress, inflammatory vascular changes, excess salt and water load. Important cofactors for the increased mortality in dialysis patients are an inadequate removal of the "uremia toxins" or a uremia-induced malnutrition.

   In patients with end-stage dialysis-dependent renal failure, increased calcification of the coronary vessels, of the cardiac valves and other myocardial tissue, as well as an increase in the calcium x phosphate product is frequently seen. An association is also seen with an increased mortality. Block and colleagues were able to show that the relative mortality risk in patients with an increased calcium x phosphate product is increased and that increased cardiovascular causes of death could be seen. An increased calcium x phosphate product potentiates the calcification of arterial vascular walls and thus produces reduced elasticity. Using electron beam computer tomography it could be shown that calcification in the region of the coronary vessels was observed much more frequently in patients with end-stage renal failure than in healthy control persons.

   In the general population it has been shown that calcium channel blockers are very good vasodilators and antihypertensive drugs. In the general population calcium antagonists of the types long-acting dihydropyridines, verapamil or diltiazem are used preferentially for the treatment of elderly patients or patients with isolated systolic hypertension. However, patients with end-stage renal failure also profit from the administration of calcium channel blockers, as these reduce the blood pressure, reduce the uremia toxin-induced calcinosis of the vessels and produce a reduced influx of calcium into the vessel walls. Calcium channel blockers inhibit macrophage proliferation. Calcium channel blockers can also reduce raised calcium levels in B-lymphocytes of patients with end-stage renal failure.

   In a preliminary retrospective investigation, the study directors investigated the effects of the administration of calcium antagonists on mortality. 188 patients with end-stage renal failure and chronic regular haemodialysis were observed for 30 months from July 1998. Parameters such as age, sex, laboratory values, clinical data and dialysis dose were recorded. Up to December 2000 51 patients had died (27%). The investigation showed advanced age and low body-mass index to be causes of increased mortality. In contrast, the availability of calcium channel blockers was favorable. After statistical analysis of the data using a Cox risk-regression model it was found that the patients taking the calcium channel blockers showed a significantly lower mortality (relative risk 0.22 [95% confidence interval 0.17-0.67] p < 0.001). This preliminary investigation thus shows that the use of calcium channel blockers significantly lowers mortality in patients with end-stage dialysis-dependent renal failure who have an increased mortality due to cardiovascular events.

   2 Ethical Aspects:

   Patients with end-stage renal failure and existing, or a history of known, arterial hypertension have a clearly increased mortality because of cardiovascular events in comparison with a normal population. So far there are no medicaments that have been demonstrated in studies to reduce the mortality of patients with dialysis-dependent renal failure. In a preliminary study there were indications that calcium channel blockers, and in particular amlodipine, lead to a reduction of cardiovascular mortality.

   The investigation will be carried out after appropriate explanation has been given and written informed consent has been obtained from the patients.

   Provisions for Monitoring of the Study by the Ethics Committee:

   The applicants, Prof. Dr. med. M. Tepel and Dr. med. M. van der Giet, are prepared to enable authorized members of the Ethics Committee to observe the trial at any time.

   3 Study Timetable:

   3.1 Justification of the Timetable: Every patient will be observed for a period of 30 months. Patients with end-stage renal failure of non-diabetic origin have a five-year survival expectation of about 35 - 40%, whereas patients with end-stage renal failure of diabetic origin have a five-year survival rate of about 20% (United States Renal Data System: Annual Data Report 2000. Am. J. Kidney Dis. 2000; 36 Suppl. 2, p. 127). It is therefore to be assumed that within 30 months about 35 - 40% of the examined patients will die. This period should be sufficient to observe any possible positive effects of amlodipine on mortality.

   The medicinal preparation is licensed for long-term therapy, so that negative effects due to the medicament are not to be expected.

   4. General Planning:

   A randomized, double-blind, placebo-controlled, multicenter study with two groups will be carried out in order to show reduction of the mortality in patients with end-stage renal failure. The study will be carried out over a period of 30 months. A check will be made every six months to see if an event has occurred.

   All patients who fulfil the inclusion criteria and who are prepared to participate in the study will be randomly assigned at the first issue of the study medicament to one of the groups. The patient will receive either amlodipine 10 mg or placebo. Both medicaments will be given as a single daily dose in the form of tablets in the morning. The study medication will not be changed during the course of the study, insofar as no side-effects are observed. Patients who are already taking a calcium channel blocker, and in whom a withdrawal phase is possible according to the opinion of their physician, will first undergo a wash-out phase of 4 weeks before starting with the double-blind treatment. During the study, the administration of all other necessary medicaments for the patient, apart from the administration of calcium channel blockers, is permitted. A check will be carried out at intervals of 6 months to see whether an event has occurred. Each patient will be observed for a period of 30 months.

   4.2 Course of the Study:

   Visit 1 (initial examination): First of all the patient will be informed about the study. If the patient consents to participate, a short clinical history and physical examination will be carried out. Then the criteria of inclusion and exclusion will be checked. The blood pressure, pulse rate and body mass index will be determined. Subsequently the patient will be asked about previous diseases, with specific questioning about the occurrence of diabetes mellitus, coronary heart disease, stroke (including transitory ischaemic attacks [TIA] and prolonged reversible ischaemic neurological deficit [PRIND]) and peripheral arterial occlusive disease. The patient will be enrolled in the study if he/she fulfils the inclusion criteria and there are no exclusion criteria. Should the patient be taking a calcium channel blocker at the time of enrolment in the study, this will be withdrawn insofar as the attending physician considers that this is possible. Other existing medication will be retained. The interval between Visit 1 and Visit 2 is one week.

   Visit 2 (start of study, month 0): The patient's current medication will be recorded (with particular reference to the following concomitant medication: ACE inhibitors, AngII blockers, statins, erythropoietin, beta-blockers). Questions will be asked about newly developed diseases with special attention to the occurrence of diabetes mellitus, coronary heart disease, stroke (including transitory ischaemic attacks [TIA] and prolonged reversible ischaemic neurological deficit [PRIND]) and peripheral arterial occlusive disease. The blood pressure, pulse rate and body mass index will be recorded. Study medication for 28 weeks will be issued. The patient will be informed about taking the medicament. Laboratory values will be recorded in the course of the routine monitoring of the patients (abbreviated and extensive routine laboratory examinations: hemoglobin, leukocyte count, platelet count, calcium, calcium x phosphate product, urea, serum creatinine, total protein, parathyroid hormone, cholesterol, triglycerides and ferritin). The patient will be asked about current symptoms.

   Visits 3 - 6 (follow-up observation, months 6, 12, 18 and 24): The current medication of the patient will be recorded (with especial emphasis on the following concomitant medications: ACE inhibitors, AngII blockers, statins, erythropoietin, beta-blockers). Questions will be asked about newly developed diseases with special attention to the occurrence of diabetes mellitus, coronary heart disease, stroke (including transitory ischaemic attacks [TIA] and prolonged reversible ischaemic neurological deficits [PRIND]) and peripheral arterial occlusive disease. The blood pressure, pulse rate and body mass index will be recorded. The study medication will be counted. New supplies of study medication for 28 weeks will be issued. Questions will be asked about side-effects. The patient will be asked about current symptoms. Laboratory values will be recorded in the course of the routine monitoring of the patient (abbreviated routine laboratory: hemoglobin, leukocyte count, platelet count, calcium, calcium x phosphate product, urea, serum creatinine, total protein).

   Visit 7 (study closure, month 30): The current medication of the patient will be recorded (with especial emphasis on the following concomitant medications: ACE inhibitors, AngII blockers, statins, erythropoietin, beta-blockers). Questions will be asked about newly developed diseases with special attention to the occurrence of diabetes mellitus, coronary heart disease, stroke (including transitory ischaemic attacks [TIA] and prolonged reversible ischaemic neurological deficits [PRIND]) and peripheral arterial occlusive disease. The blood pressure, pulse rate and body mass index will be recorded. The study medication will be counted. Questions will be asked about side-effects. The patient will be asked about current symptoms. Laboratory values will be recorded in the course of the routine monitoring of the patients (abbreviated and extensive routine laboratory: hemoglobin, leukocyte count, platelet count, calcium, calcium x phosphate product, urea, serum creatinine, total protein, parathyroid hormone, cholesterol, triglycerides and ferritin).

   After completing the study, the data will be recorded after unblinding and evaluated (duration about 2 months) and prepared for publication.

   Checks on the Observation of the Protocol: The study directors will employ a monitor for the duration of the study who will visit all the centers at intervals of six months and check observation of the study protocol.

   4.3 Study Medication (trial preparation, blinding, concomitant medication):

   Amlodipine 10 mg will be used as the trial preparation Amlodipine is a calcium antagonist that has already been the licensed within the European Union for the indications: essential hypertension, chronic stable angina pectoris (angina on effort). Placebo will be used as control.

   4.3.1 Blinding:

   All members of the study team and all personnel who are involved in the course of the study will work under blind conditions throughout the entire period of the trial. The study directors and investigators will be provided with the randomization code in sealed envelopes. The placebo and active drug do not differ in form, color, odor or weight.

   4.3.2 Actions and Unblinding for Side-Effects:

   Blinding is essential in order to maintain the integrity of the study. Should, however, an emergency develop in which knowledge of the substance administered is necessary, then the blinding can be broken by the attending physician. If unblinding takes place, the responsible study directors must be contacted. All cases of unblinding will be recorded in the study record sheets. The study directors may be contacted in emergencies at any time by the telephone hotline (+ 49-30 8445 2305). Reports on serious adverse events should be made within 24 hours. These reports of serious adverse events must be sent to the study directors (Prof. Dr. med. M. Tepel or Dr. med. van der Giet, Freie Universität Berlin, Universitätsklinikum Benjamin Franklin, Medizinische Klinik IV, Hindenburgdamm 30, 12200 Berlin, Tel/Fax: +49-30 8445 2305). Other side-effects will be recorded by the attending physician, documented and registered at the control visits.

   4.3.3 Concomitant Medication:

   The patients may take all the medicines that their attending physicians consider to be necessary throughout the course of the study. Exception: the administration of a calcium channel blocker during the study is not permissible. The medication will be recorded in detail at the regular monitoring visits.

   5. Objectives:

   5.1 Primary Parameters: The primary parameter will be the survival rate.

   5.2 Secondary Parameters: No secondary parameters will be investigated during the study.

   5.3 Methods for Recording Efficacy and Safety:

   All patients will be encouraged to maintain their diet and regular physical exercise throughout the duration of the study.

   All patients will be followed up at intervals of 6 months. At these visits, side-effects and changes in vital status will be recorded.

   When the medicament is issued for the first time, all patients will be observed for 2 hours after taking it.

   5.4 Compliance: The study medication and the concomitant medicaments will be checked at 6 month intervals. If necessary, the patients will be reminded of the necessity to take the drug.

   6. Data Management: All data for the study will be entered in the Clinical Record Forms and submitted for central analysis of the data (study directors). One copy of the Clinical Record Form will be retained by the attending physician. The study directors will ensure that the data are analyzed and statistically evaluated. Current Data Protection Regulations will be observed. The data will be analyzed in an anonymised form. The patient must consent to the data being recorded in the context of the clinical trial, being analyzed and being submitted at the request of the pertinent supervisory authorities. Each patient will be assigned a number on enrolment in the study and his /her initials will be recorded. Unequivocal patient identification will be possible via a patient identification list consisting of the patient number, initials, date of birth, name and first name. All data will be archived for a period of 10 years.

   6.1 Statistical Procedures:

   This 30-month-long, double-blind, placebo-control study is intended to show that the administration of calcium antagonists reduces the mortality of patients undergoing regular haemodialysis.

   The hypotheses to be tested are:

   H0: the mortality rates are the same; HA: the mortality rates are different.

   The log-rank test will be used to test for possible statistically significant differences (probability p = 0.05, two-tailed test).

   It is not intended to carry out any interim analysis.

   6.2 Estimation of Number of Cases:

   The sample size is calculated by comparison of two survival curves (Computer-Programm: "n-Query": Log-rank-Test of survival in two groups).

   The size of the sample is calculated on the basis of alpha = 0.05, power 80%, two-tailed test for a difference of 14% between amlodipine and placebo with a sample size of 163 per group (log-rank test or survival in two groups, followed for fixed time, constant hazard ratio). Expected mortality rate: placebo 40% and amlodipine 26% .

   It is assumed that 30 patients will drop out of the study from the two groups together (e.g. change of dialysis center).

   Therefore, 356 patients (178 patients amlodipine versus 178 patients placebo) are to be investigated.

   7. Financing of the Study:

   The study will be supported financially and materially by the Pfizer company (Karlsruhe). The company will provide the medication/placebo.

   8. Miscellaneous:

   8.1 Insurance and Liability:

   An application for patient insurance has been made to the Gerling company and will be accordingly submitted.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease
* Hemodialysis
* Hypertension
* Written informed consent

Exclusion Criteria:

* Hypotension of less than 90 mmHg systolic
* High-grade aortic stenosis
* Heart failure of NYHA stage III and IV
* Acute myocardial infarction (within the last 4 weeks)
* Acute heart failure
* Known allergy to the medicament amlodipine or other constituents of the medicament
* Severe disorders of liver function
* Pregnancy and breast-feeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2002-01; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the survival rate. The secondary outcome will be cardiovascular events. | Prospective: look forward using periodic observations collected predominantly following subject enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Martin Tepel, Dr, Principal Investigator — Charite Campus Benjamin Franklin
Locations (1):
- Charite Campus Benjamin Franklin, Berlin, Germany

REFERENCES:
- [Background] Tepel M, Giet MV, Park A, Zidek W. Association of calcium channel blockers and mortality in haemodialysis patients. Clin Sci (Lond). 2002 Nov;103(5):511-5. doi: 10.1042/cs1030511. PMID 12401125
- [Derived] Mugendi GA, Mutua FM, Natale P, Esterhuizen TM, Strippoli GF. Calcium channel blockers for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 Oct 1;10(10):CD011064. doi: 10.1002/14651858.CD011064.pub2. PMID 33000470
- [Derived] Tepel M, Hopfenmueller W, Scholze A, Maier A, Zidek W. Effect of amlodipine on cardiovascular events in hypertensive haemodialysis patients. Nephrol Dial Transplant. 2008 Nov;23(11):3605-12. doi: 10.1093/ndt/gfn304. Epub 2008 May 29. PMID 18511605